CLINICAL TRIAL: NCT06358443
Title: The Long-term Effect on Bone Markers (BM) and Body Mineral Density (BMD) of Daily Jarlsberg Cheese Intake in Patient With Osteopenia
Brief Title: The Long-term Effect of Daily Jarlsberg Cheese Intake in Patient With Osteopenia
Acronym: PF-JB3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Tine (Industry)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PF-Jarlsberg/IIIB
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Osteopenia; Osteoporosis
Keywords: Jarlsberg cheese; BMD; BTM; Osteocalcin
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Calcium

STUDY DESIGN:
Intervention Model Description: One armed observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jarlsberg cheese + vitamin D and Calcium tablets (Experimental): All the patients will receive optimal daily efficacy dose of Jarlsberg cheese pluss vitamin D ampulles and calcium tablets in one year
  Interventions: Dietary Supplement: Jarlsberg cheese

INTERVENTIONS:
Dietary Supplement: Jarlsberg cheese — Jarlsberg cheese + Vitamin D ampulles + Calcium
  Other Names: Vitamin D ampulles; Calcium tablets

SUMMARY:
Aim: To estimate the effect of daily optimal efficacy dose (OED) of Jarlsberg cheese in patients with Osteopeni (OP).

Study population: Post-menopausal women and men above 55 years of age in risk of Osteoporosis Treatment: Daily OED Jarlsberg cheese + vitamin D and Calcium tablets. Design: An open and one-armed observational study. Main variables: Bone Mineral Density (BMD), Bone turnover markers (BTMs), Osteocalcin and K2 vitameres.

Study Procedure: Prior to inclusion in this study, all the patients have undergone 32 days of daily OED intake of Jarlsberg cheese + vitamin D and caicium tablets. Thid is the baseline of this observational study. The duration of this study is 12 months with clinical examination and bloodsampling after 6 and 12 months.

Sample size: At least 16 patients will be included

DETAILED DESCRIPTION:
Aim: To estimate the short- and long-term effect of daily optimal efficacy dose (OED) of Jarlsberg cheese on BMD, bone turn-over markers (BTMs) and Osteocalcin in patients with Osteopeni (OP).

Study population: The study population consists of OP-patients of post-menopausal women and men above 55 years of age who had a daily OED intake of Jarlsberg Cheese 32 weeks prior to inclusion in the study. OP patients are defined as patients with a T-score below 0.0 but larger than -2.5.

Trial treatment: The optimal daily intake of Jarlsberg cheese depending on gender, age, and physical activity. Women in post-menopausal age have a daily OED Jarlsberg of 47gram and men in above 55 years of age have an estimated daily OED of 71gram.The cheese will be delivered in package of 250 gram with slices average of 15.625gram. 47 gram represents 3 slices and 67 gram 4.5 slices. In addition to Jarlsberg Cheese, all the included patients will receive 40mcg vitamin D and 500 mg Ca.

Design: The study will be performed as a follow-up study of a randomized, single-blinded Norwegian multicentre trial with stratified semi-cross-over design with gender and participating General Practitioner (GP) site as stratification factors. GP's from Viken county will participate. This follow-up part will be performed as an open and one-armed observational study.

Main variables: The main response variable will be the change in Bone Mineral Density (BMD) and recorded at baseline follow-up after 32 weeks with daily Jarlsberg intake and the end of the follow-up study (Week 52). The second main variables will be total Osteocalcin (tOC), carboxylated osteocalcin (cOC), the osteocalcin ratio RO defined as the ratio between cOC and under-carboxylated osteocalcin (ucOC) [RO = cOC / ucOC] recorded at baseline-FU, week 26 and week 52. Additionally, the bone turnover markers (BTMs) cross-linked C-telopeptide type I collagen (CTX), procollagen type 1 N-terminal propeptide (PINP), bone specific ALP (BALB) and Parathyroid hormone (PTH) will be measured at the same visits. At baseline-FU and week 52, the following variables will be measured: Vitamin K2 and the different vitamers MK-7, MK-8, MK-9, and MK-9(4H) used as explanatory variable, Diet registration as controlling variables and HbA1C, Lipids, biochemical variables together with "Quality-of-Life" (QoL) questionnaire as supporting variables. The Interleukins IL-1β, IL6, IL8, IL10 and the Cytokines TNF-α, NF-ƙβ (RANK-L), OPG and TGF-β will be measured at baseline-FU and at the last visit in the study (Week 52). The Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) will be used for registration of Adverse Events (AE) and toxicity score at all investigation visits.

Study procedure

Baseline of Follow-up: Patients who completed 32 weeks of daily intake of Jarlsberg OED in the PF-Jarlsberg/IIIA and willing to give informed consent to participate in the follow-up part will be included. The baseline for the follow-up part will be the last control in the PF-Jarlsberg/IIIA. This includes measurements of BMD, Osteocalcin, CTX-1, PINP, BALP, PTH and vitamin K. Additionally, blood samples for measuring of the central biochemical variables and registration of the food intake during four consecutive days will be performed. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 used for measuring and classifying the tolerability and toxicity will be recorded as well. The included patients will receive Jarlsberg Cheese, vitamin D- and Ca tablets as in the previous study for eight weeks. The daily intake of Jarlsberg will be 47gram for women and 71gram for men, combined with 40μg vitamin D and 500 mg Ca. The patients will be given a Compliance & Activity form (CAF) and asked to write down the daily intake of treatment medicine, Jarlsberg cheese and hours of physical activities.

Clinical part: All the participants will get a new delivery Jarlsberg Cheese, vitamin D and Ca-tablets every eight weeks. The patients will return the CAF for the previous period and receive a new CAF to fill in every day during the next eight-week period. After 26 weeks in the Follow-up, the patients meet for a new visit at the Medical Centre. At this visit a physical examination will be performed, blood samples for measurement of Osteocalcin, CTX-1, PINP, BALP, PTH and the central biochemical variables will be taken, concomitant medication and treatment compliance recorded.

The participating patients will receive Jarlsberg, vitamin and Ca-tablets at week 8,16, 24, 32, 40 and 48. The final visit and physical examination in the Follow-up study will be performed at week 52. This includes measurements of BMD, Osteocalcin, BTMs and vitamin K. Additionally, blood samples for measuring lipides, HbA1C and the central biochemical variables and registration of the daily food intake during four consecutive days will be performed. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 used for measuring and classifying the tolerability and toxicity will be recorded as well.

Sample size: The change from baseline FU to week 52 in BMD expressed by the 95% Confidence Interval of the change must be ≤ SD in change of BMD, at least 16 patients in each gender group must finalize the study.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women and men passed the age of 55 years suffering from Osteopeni and had a daily Optimal Effective Dose of Jarlsberg Cheese the last 32 weeks prior to inclusion.

Exclusion Criteria:

* • Diagnosed eating disorder.

  * Serious gastrointestinal disorder.
  * Serious liver or kidney disease. (GFR<29 mL/min/1,73m2)
  * Diabetes mellitus type I.
  * Diabetes type II without sufficient control.
  * Suffering from verified cancer.
  * Under systemic treatment with corticosteroids the last 3 weeks before start of the trial treatment.
  * Under active antiresorptive treatment or anabolic treatment.
  * Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment except from Jarlsberg cheese .
  * Known milk protein allergy.
  * Not able to understand information.
  * Do not want or not able to give written consent to participate in the study.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Baseline, 6 months, 12 months
  Bone health
Bone Turnover Markers | Baseline, 6 month, 12 months
  Bone health
Osteocalcin | Baseline, 6 month, 12 months
  Bone health

SECONDARY OUTCOMES:
Vitamin K2 | Baseline, 6 month, 12 months
  K2 vitameres

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Whist, PhD, Study Director — Tine
Locations (1):
- Skjetten Medical center, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No